CLINICAL TRIAL: NCT07045142
Title: Metformin Alleviates Abnormal Glucose Metabolism Induced by Statins in Schizophrenia Patients: A Randomized, Double-Blind, Placebo-Controlled Multicenter Clinical Study
Brief Title: Metformin Alleviates Abnormal Glucose Metabolism Induced by Statins in Schizophrenia Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Central South University (Other)
Collaborators: Zhumadian Second People's Hospital (Unknown); The Third Hospital of Changsha County (Unknown); The Second People's Hospital of Dali Bai Autonomous Prefecture (Unknown); Xiangshan County Traditional Chinese Medicine Hospital Medical and Health Group Three Hospitals Distric (Unknown); Yueyang Rehabilitation Hospital (Unknown)
Responsible Party: Principal Investigator, Renrong Wu, Professor, Central South University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: WU202505STA
Record Dates: First submitted 2025-06-22; First posted 2025-07-01 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-07

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Dyslipidemia; Metformin; Statin
MeSH Terms: conditions — Schizophrenia; Dyslipidemias | interventions — Atorvastatin; Metformin

STUDY DESIGN:
Intervention Model Description: We will include 200-400 schizophrenia patients with dyslipidemia from the Second Xiangya Hospital and other sites, randomly assigning them to receive either atorvastatin with metformin or atorvastatin with placebo. Two groups were observed longitudinally for 6 months.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin group (Active Comparator): To explore the impact of metformin on glucose metabolism abnormalities in schizophrenia patients undergoing atorvastatin treatment.
  Interventions: Drug: Atorvastatin; Drug: Metformin
- Placebo group (Placebo Comparator): To serve as a placebo control for evaluating the effects of atorvastatin treatment on glucose metabolism in schizophrenia patients, isolating the impact of metformin from the effects of atorvastatin.
  Interventions: Drug: Atorvastatin; Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin — Participants will receive atorvastatin 20 mg daily.
Drug: Metformin — Participants will receive metformin 1000 mg daily.
  Arms: Metformin group
Drug: Placebo — Participants will receive placebo 1000 mg daily, mimicking the appearance of metformin without containing active ingredients.
  Arms: Placebo group

SUMMARY:
Schizophrenia is a severe mental illness associated with significant morbidity and disability. Patients often experience metabolic side effects from antipsychotic medications, including weight gain and dyslipidemia. Statins, commonly used to manage dyslipidemia, can lower cholesterol levels but may increase the risk of new-onset diabetes.

This study aims to investigate how atorvastatin affects glucose metabolism in schizophrenia patients and assess whether metformin can help improve these metabolic issues. The investigators will include 200 patients with dyslipidemia from the Second Xiangya Hospital and other sites, randomly assigning them to receive either atorvastatin with metformin or atorvastatin with placebo over six months.

Key goals include evaluating the impact of atorvastatin on insulin resistance and blood glucose levels and determining the effectiveness of metformin in mitigating glucose metabolism abnormalities while managing lipid levels.

Understanding these interactions will help improve treatment strategies for schizophrenia patients, potentially lowering their risk of cardiovascular diseases and diabetes and enhancing overall health outcomes.

DETAILED DESCRIPTION:
Research Background: Schizophrenia is a severe mental disorder characterized by high morbidity, significant disability, and substantial disease burden. Studies have shown that antipsychotic medications, particularly atypical antipsychotics, can lead to considerable metabolic side effects, including weight gain, hyperlipidemia, hyperglycemia, and insulin resistance. Statins are widely used for cardiovascular disease prevention and treatment in high-risk populations. Schizophrenia patients are at an increased risk of dyslipidemia due to long-term antipsychotic medication use, with research indicating that approximately 66% of chronic schizophrenia patients develop varying degrees of dyslipidemia following antipsychotic treatment. Dyslipidemia not only accelerates cardiovascular disease progression but may also lead to premature mortality, with schizophrenia patients facing double the risk of cardiovascular death compared to the general population, resulting in a reduction of lifespan by 9 to 12 years. As such, monitoring and intervening in dyslipidemia among these patients are crucial for improving long-term prognosis. However, while long-term statin use can mitigate myocardial infarction risk, it also raises the risk of new-onset diabetes, with evidence suggesting a 10% increase in diabetes risk attributable to statins-a factor that has not been thoroughly examined in the context of glucose metabolism in schizophrenia patients.

Research Objective: This study aims to explore the occurrence of glucose metabolism abnormalities in schizophrenia patients undergoing atorvastatin treatment for dyslipidemia and to evaluate the ameliorative effects of metformin. Specific objectives include: 1) Investigating the impact of atorvastatin on glucose metabolism by observing changes in insulin resistance, fasting blood glucose, and glycated hemoglobin levels to assess atorvastatin's potential effects on glucose metabolism; 2) Evaluating the adjunctive role of metformin by randomly assigning eligible patients to either a metformin treatment group or a placebo group to observe the auxiliary effect of metformin in atorvastatin therapy and assess its impact on glucose metabolism abnormalities and underlying mechanisms; and 3) Examining the metabolic effects of metformin on dyslipidemia by assessing its influence on lipid profiles (e.g., LDL-C, total cholesterol, triglycerides) during atorvastatin treatment while controlling for glucose metabolism abnormalities.

Research Plan: This study will recruit 200 schizophrenia patients from the Second Xiangya Hospital of Central South University and other partnering institutions. Eligible participants must be aged 18 to 65, meet the criteria for schizophrenia, have stable symptoms and medication regimens for over three months. Participants will provide informed consent prior to inclusion. For lipid levels, participants must meet at least one of the following criteria: 1) fasting total cholesterol (TC) ≥ 5.2 mmol/L; 2) fasting triglycerides (TG) ≥ 1.7 mmol/L; 3) fasting low-density lipoprotein cholesterol (LDL-C) ≥ 3.4 mmol/L. For blood glucose, participants must have two consecutive fasting blood glucose (FPG) tests < 6.1 mmol/L, with an interval of 1-4 weeks between tests. Patients with a prior diagnosis of diabetes, diabetic ketoacidosis, or any other diabetes-related complications are excluded. Participants will provide informed consent prior to inclusion. The study employs a randomized controlled trial (RCT) design, with participants randomly assigned to two groups: one group receiving atorvastatin 20 mg/day combined with metformin 1000 mg/day and the other receiving atorvastatin 20 mg/day with a placebo. The study duration is six months, with follow-ups at 3 and 6 months, including baseline assessments and multiple blood tests to monitor glucose metabolism and other relevant indices.

Expected Outcomes: By evaluating the effects of atorvastatin on glucose metabolism in schizophrenia patients and the intervention effects of metformin, this study seeks to elucidate the risk of glucose metabolism abnormalities associated with statin therapy in this population and the mechanisms through which metformin improves these outcomes. This research will contribute to developing more effective treatment regimens for schizophrenia patients, thereby reducing cardiovascular disease and diabetes risks and improving patient prognosis. Additionally, results may facilitate the integration of management practices for both mental and metabolic disorders, reducing the healthcare burden from metabolic complications.

ELIGIBILITY:
Inclusion criteria:

1. Aged between 18 and 65 years, regardless of gender, and meets the diagnostic criteria for schizophrenia according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5);
2. Symptoms and medication regimen stable for more than 3 months, with the allowance of up to two antipsychotic medications in combination (concurrent use of antidepressants, anxiolytics, and mood stabilizers is permitted);
3. Temporary use of benzodiazepines is allowed;
4. Meets at least one of the following conditions: fasting total cholesterol (TC) ≥ 5.2 mmol/L; fasting triglycerides (TG) ≥ 1.7 mmol/L; fasting low-density lipoprotein cholesterol (LDL-C) ≥ 3.4 mmol/L;
5. Two fasting blood glucose (FPG) tests must be < 6.1 mmol/L (with an interval of 1-4 weeks);
6. It is anticipated that there will be no issues related to relocation, transportation difficulties, or access to medical care throughout the study;
7. Informed consent must be obtained from the patient and their guardian, and a consent form must be signed.

Exclusion criteria:

1. Patients with a prior diagnosis of diabetes or complications such as diabetic ketoacidosis;
2. Patients with liver or kidney dysfunction, indicated by aspartate aminotransferase (AST), alanine aminotransferase (ALT), or gamma-glutamyl transferase (GGT) levels exceeding twice the normal limits, and/or creatinine levels exceeding 1.2 times the upper limit of the reference range or greater than 2 mg/dL, or deemed by the investigator to have liver and/or kidney impairment that warrants exclusion from the study;
3. Patients with severe gastrointestinal, respiratory, endocrine, hematologic diseases, or metabolic absorption disorders: including but not limited to poorly controlled diabetes, severe acute systemic infections or immunological diseases, ischemic heart disease, cerebrovascular accidents within the past year, history of prolonged QT interval, active hepatitis B virus, chronic active hepatitis C, and malabsorption syndromes;
4. Clinically significant abnormal ECG findings at screening that the investigator deems unsuitable for inclusion, such as male QTc interval > 470 ms, female QTc interval > 480 ms;
5. Pregnant or nursing women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Fasting Blood Glucose Concentration | Baseline, 3rd month, 6th month
Change from Baseline in Glycated Hemoglobin (HbA1c) Concentration | Baseline, 3rd month, 6th month
Oral Glucose Tolerance Test | Baseline, 3rd month, 6th month
  The Oral Glucose Tolerance Test (OGTT) requires subjects to undergo an 8-hour fasting period, followed by an initial measurement of fasting blood glucose via a portable glucometer using a finger prick. Subsequently, subjects are instructed to consume a solution containing 75 grams of anhydrous glucose dissolved in 300 milliliters of water. Blood samples are then collected through finger pricking at 1 hour and 2 hours post-ingestion for further analysis of glucose levels.

SECONDARY OUTCOMES:
Change from Baseline in Fasting insulin Concentration | Baseline, 3rd month, 6th month
Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) | Baseline, 3rd month, 6th month
  HOMA-IR (Homeostasis Model Assessment of Insulin Resistance) is a recognized method for estimating insulin resistance, which plays a critical role in metabolic disorders such as type 2 diabetes and cardiovascular disease. This assessment requires fasting for at least eight hours, followed by the measurement of fasting insulin and fasting glucose levels from blood samples. The HOMA-IR value indicates the degree of insulin resistance; higher values suggest reduced cellular responsiveness to insulin, thereby correlating with increased risk for metabolic syndrome and type 2 diabetes.
Change from Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score | Baseline, 3rd month, 6th month
  Range: 30 to 210; Higher Scores Indicate Worse Symptoms.
Change from Baseline in Global Assessment of Functioning Scale (GAF) Total Score | Baseline, 3rd month, 6th month
  Range: 0 to 100; Higher Scores Indicate Better Functioning.
Abdominal ultrasound examination. | baseline, 6 months
  Abdominal ultrasound is performed only at designated study sites and serves as a secondary outcome.The abdominal ultrasound examination will focus on assessing the occurrence of metabolic associated fatty liver disease (MAFLD). Subjects are required to fast for at least 8 hours prior to the examination, and they will lie supine on the examination table. After applying a coupling agent, an ultrasound scan will be performed. The physician will measure the size of the liver, observe its echo characteristics, and assess the echo differences with surrounding organs to determine the presence of liver enlargement or fat deposition. MAFLD typically presents as increased hepatic echogenicity and blurred liver margins. Doppler ultrasound may also be used to evaluate hepatic blood flow if necessary. All examination results will be recorded on case report forms for comprehensive analysis to assess the metabolic status and the degree of MAFLD in the study subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Renrong Wu, Study Chair — Mental Health Institute of Second Xiangya Hospital,CSU
Locations (6):
- China (6):
  - Zhumadian Second People's Hospital, Zhumadian, Henan
  - Mental Health Institute of Second Xiangya Hospital, CSU, Changsha, Hunan
  - The Third Hospital of Changsha County, Changsha, Hunan
  - Yueyang Rehabilitation Hospital, Yueyang, Hunan
  - The Second People's Hospital of Dali Bai Autonomous Prefecture, Dali, Yunnan
  - Xiangshan County Traditional Chinese Medicine Hospital Medical and Health Group Three Hospitals District, Xiangshan, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Result] Sasaki J, Otonari T, Uchida Y, Ikeda Y, Biro S, Kono S; PRAT study investigators. Effects of pravastatin and atorvastatin on HDL cholesterol and glucose metabolism in patients with dyslipidemia and glucose intolerance: the PRAT study. J Atheroscler Thromb. 2013;20(4):368-79. doi: 10.5551/jat.13532. Epub 2012 Dec 15. PMID 23257975
- [Result] Preiss D, Seshasai SR, Welsh P, Murphy SA, Ho JE, Waters DD, DeMicco DA, Barter P, Cannon CP, Sabatine MS, Braunwald E, Kastelein JJ, de Lemos JA, Blazing MA, Pedersen TR, Tikkanen MJ, Sattar N, Ray KK. Risk of incident diabetes with intensive-dose compared with moderate-dose statin therapy: a meta-analysis. JAMA. 2011 Jun 22;305(24):2556-64. doi: 10.1001/jama.2011.860. PMID 21693744
- [Result] Sattar N, Preiss D, Murray HM, Welsh P, Buckley BM, de Craen AJ, Seshasai SR, McMurray JJ, Freeman DJ, Jukema JW, Macfarlane PW, Packard CJ, Stott DJ, Westendorp RG, Shepherd J, Davis BR, Pressel SL, Marchioli R, Marfisi RM, Maggioni AP, Tavazzi L, Tognoni G, Kjekshus J, Pedersen TR, Cook TJ, Gotto AM, Clearfield MB, Downs JR, Nakamura H, Ohashi Y, Mizuno K, Ray KK, Ford I. Statins and risk of incident diabetes: a collaborative meta-analysis of randomised statin trials. Lancet. 2010 Feb 27;375(9716):735-42. doi: 10.1016/S0140-6736(09)61965-6. Epub 2010 Feb 16. PMID 20167359
- [Result] Pillinger T, McCutcheon RA, Vano L, Mizuno Y, Arumuham A, Hindley G, Beck K, Natesan S, Efthimiou O, Cipriani A, Howes OD. Comparative effects of 18 antipsychotics on metabolic function in patients with schizophrenia, predictors of metabolic dysregulation, and association with psychopathology: a systematic review and network meta-analysis. Lancet Psychiatry. 2020 Jan;7(1):64-77. doi: 10.1016/S2215-0366(19)30416-X. Epub 2019 Dec 17. PMID 31860457